CLINICAL TRIAL: NCT00099268
Title: A Long Term, Double-blind, Randomized, Parallel-group, Carbidopa/Levodopa Controlled, Multi-center Study to Evaluate the Effect of Carbidopa/Levodopa/Entacapone in Patients With Parkinson's Disease Requiring Initiation of Levodopa Therapy
Brief Title: Efficacy and Safety of Carbidopa/Levodopa/Entacapone in Patients With Parkinson's Disease Requiring Initiation of Levodopa Therapy
Acronym: STRIDE-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CELC200A2401
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, levodopa therapy, dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Stalevo; Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Carbidopa/levodopa/entacapone (Experimental): Patients received Carbidopa/levodopa/entacapone tablets. The study was designed as a flexible dose trial (200-1000 mg/day levodopa). The target dose was 400 mg/day levodopa administered orally as 4 equal doses 4 times a day with 3.5-hour dosing intervals for a treatment period of 134 to 208 weeks.
  Interventions: Drug: Carbidopa/levodopa/entacapone
- Immediate release carbidopa/levodopa (Active Comparator): Patients received Immediate release carbidopa/levodopa tablets. The study was designed as a flexible dose trial (200-1000 mg/day levodopa). The target dose was 400 mg/day levodopa administered orally as 4 equal doses 4 times a day with 3.5-hour dosing intervals for a treatment period of 134 to 208 weeks.
  Interventions: Drug: Immediate release carbidopa/levodopa

INTERVENTIONS:
Drug: Carbidopa/levodopa/entacapone — Carbidopa/Levodopa/Entacapone 12.5/50/200 mg and 25/100/200 mg capsules.
  Other Names: Stalevo
  Arms: Carbidopa/levodopa/entacapone
Drug: Immediate release carbidopa/levodopa — Immediate release carbidopa/levodopa 12.5/50 mg and 25/100 mg capsules.
  Other Names: Sinemet
  Arms: Immediate release carbidopa/levodopa

SUMMARY:
The CELC200A2401 study has been designed in order to evaluate the hypothesis that administering the combination carbidopa/levodopa/entacapone at the time that levodopa therapy is initiated results in a decrease in the risk of the development of motor complications for patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease
* Diagnosis of Parkinson's disease for no more than 5 years

Exclusion Criteria:

* History, signs, or symptoms of atypical or secondary parkinsonism
* Presence at baseline of drug-related wearing-off symptoms, dyskinesia or other motor complications
* Levodopa exposure of more than 30 days or anytime within 8 weeks prior to visit 1

Other inclusion/exclusion criteria applied to this study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2004-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Coastal Neurological Medical Group, La Jolla, California
  - Keck School of Medicine, Division of Movement Disorders, Los Angeles, California
  - Reed Neurological Research Center, Los Angeles, California
  - The Parkinson's Institute, Sunnyvale, California
  - Molecular NeuroImaging, LLC, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorder Center, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - Charlotte Neurological Service, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Wesley Woods Health Center, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Landon Center on Aging, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Boston University School of Medicine, Boston, Massachusetts
  - Clinical Neuroscience Center, Southfield, Michigan
  - Parkinson's Disease and Movement Disorder Center of Albany Medical, Albany, New York
  - Parkinson's Disease and Movement Disorders Center of Long Island, Commack, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, Neurological Institute, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center Movement Disorders Center, Durham, North Carolina
  - Pennsylvania Neurology Institute, Philadelphia, Pennsylvania
  - NeuroHealth, Inc., Warwick, Rhode Island
  - Semmes-Murphey Clinic, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Parkinson's Disease Center, Houston, Texas
  - Wisconsin Institute for Neurologic and Sleep Disorders, Milwaukee, Wisconsin
- Novartis Investigative Site, Innsbruck, Austria
- Belgium (2):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
- Canada (4):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Finland (5):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Mikkeli
  - Novartis Investigative Site, Oulu
  - Novartis Investigative Site, Pori
- France (4):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Tübingen
- Greece (2):
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Thessaloniki
- Italy (6):
  - Novartis Investigative Site, Catania
  - Novartis Investigative Site, Chieti Scalo
  - Novartis Investigative Site, Lido di Camaiore
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Pozzilli
  - Novartis Investigative Site, Roma
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Sweden (4):
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Norrköping
  - Novartis Investigative Site, Stockholm
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)
- United Kingdom (4):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Stocchi F, Rascol O, Kieburtz K, Poewe W, Jankovic J, Tolosa E, Barone P, Lang AE, Olanow CW. Initiating levodopa/carbidopa therapy with and without entacapone in early Parkinson disease: the STRIDE-PD study. Ann Neurol. 2010 Jul;68(1):18-27. doi: 10.1002/ana.22060. PMID 20582993

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbidopa/Levodopa: Patients received Immediate release carbidopa/levodopa tablets. The study was designed as a flexible dose trial (200-1000 mg/day levodopa). The target dose was 400 mg/day levodopa administered orally as 4 equal doses 4 times a day with 3.5-hour dosing intervals for a treatment period of 134 to 208 weeks.
Period: Overall Study
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Started | 374 | 373
Intent-to-Treat | 373 (One patient from each group discontinued without receiving a single dose of study drug.) | 372
Completed | 282 (Plus 1 death in the carbidopa/levodopa/entacapone group within 30 days of treatment discontinuation) | 291 (Plus 1 death in the carbidopa/levodopa group within 30 days of treatment discontinuation)
Not Completed | 92 | 82
Not completed — Withdrawal by Subject | 46 | 28
Not completed — Adverse Event | 19 | 19
Not completed — Protocol Violation | 9 | 8
Not completed — Lost to Follow-up | 6 | 4
Not completed — Lack of Efficacy | 5 | 18
Not completed — Administrative problems | 4 | 4
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa | Total
Number analyzed (Participants) | 373 | 372 | 745
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline numbers represent the Intent-to-treat (ITT) population. Of the 747 randomized patients, one patient in each group discontinued the study without receiving a single dose of study drug and was excluded from the ITT population.
  years | 60.6 (8.67) | 59.8 (8.20) | 60.2 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 150 | 278
  Male | 245 | 222 | 467

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Dyskinesia
Description: Dyskinesia was assessed by a blinded rater at each visit. Time to dyskinesia was defined as the visit at which the rater first answered "yes" to the following question: "In your opinion, does this patient have dyskinesia?" Time to dyskinesia was estimated by Kaplan-Meier product limit estimate that takes into consideration patients who did not experience dyskinesia by censoring them at the end of the study.
Time Frame: Treatment duration for an individual patient varied between a minimum of 134 weeks for those patients recruited last and a maximum of 208 weeks for those patients recruited first
Population: The intent to treat (ITT) population consisted of all patients randomized who received at least one dose of study drug. Following the ITT principle, patients were analyzed according to the treatment they were assigned at randomization.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Number analyzed (Participants) | 373 | 372
weeks | 90.7 (47.9) [65.3 to 104.0] | 117.1 (51.5) [92.1 to 132.6]

2. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score (Parts II and III)
Description: The UPDRS is a standardized assessment scale used to measure the patient's disease state. It was to be completed by a blinded rater. There are 6 parts to the UPDRS. Part II (items 5-17; total score 0-52 units on the scale) measures the patient's activities of daily living and part III (items 18-31; total score 0-56 units on the scale) measures the motor function of the patient. The total score ranges from 0 to 108 units on the scale. A higher score indicates greater disability. A negative change score indicates improvement.
Time Frame: Baseline, Week 6 and Week 130
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Number analyzed (Participants) | 373 | 372
Units on a scale
  Change from baseline to Week 6 | 21.9 (11.96) | 21.8 (11.24)
  Change from baseline to Week 130 | 23.2 (13.38) | 22.8 (13.21)

3. Secondary Outcome: Occurrence of Wearing-off
Description: Wearing-off is defined as a perception of loss of mobility or dexterity, usually taking place gradually over minutes (up to an hour) and usually bearing a close temporal relationship to the timing of anti-parkinsonian medications; it does not include early-morning akinesia. To ascertain its occurrence, a blinded rater questioned the patient as to whether he/she had noticed that the benefits of the study drug were wearing-off.
Time Frame: Baseline to Week 134
Population: The intent to treat (ITT) population consisted of all patients randomized who received at least one dose of study drug. Following the ITT principle, patients were analyzed according to the treatment they were assigned at randomization. Subjects who discontinued treatment before 134 weeks without wearing-off were excluded.
Measure: Number; unit: Participants
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Number analyzed (Participants) | 305 | 333
Participants | 139 (45.6) | 161 (48.3)

4. Secondary Outcome: Time to First Occurrence of Wearing-off
Description: Wearing off is defined as a perception of loss of mobility or dexterity, usually taking place gradually over minutes (up to an hour) and usually bearing a close temporal relationship to the timing of anti-parkinsonian medications; it does not include early-morning akinesia. To ascertain its occurrence, a blinded rater questioned the patient whether he/she had noticed that the benefits of the study drug wear-off. A motor complications and patient questionnaire card were provided to assist the blinded rater in determining whether a patient had experienced wearing-off.
Time Frame: Baseline to end of study (134-208 weeks of treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Weeks
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Number analyzed (Participants) | 373 | 372
Weeks | 131.7 (3.8) | 129.5 (3.6)

5. Secondary Outcome: Occurrence of Dyskinesia
Description: Dyskinesia was assessed by a blinded rater at each visit. Time to dyskinesia was defined as the visit at which the rater first answered "yes" to the following question: "In your opinion, does this patient have dyskinesia?"
Time Frame: Baseline to Week 208
Population: The intent to treat (ITT) population consisted of all patients randomized who received at least one dose of study drug. Following the ITT principle, patients were analyzed according to the treatment they were assigned at randomization. Subjects who discontinued from treatment before 134 weeks without dyskinesia were excluded.
Measure: Number; unit: Participants
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Number analyzed (Participants) | 307 | 318
Participants | 128 (41.7) | 103 (32.4)

6. Secondary Outcome: Change From Baseline in Health-related Quality of Life Assessed Using the 39-item Parkinson's Disease Questionnaire (PDQ-39)
Description: The PDQ-39 instrument is used to assess quality of life in individuals with Parkinson's disease. The questionnaire provides scores on eight scales: Mobility, activities of daily living, emotions, stigma, social support, cognition, communication, and bodily discomfort. Questions are scored on a 5-point Likert scale ranging from 1 (never) to 3 (sometimes) to 5 (always). The total score can range from 39 to 190. A lower score indicates better quality of life. A negative change score indicates an improvement.
Time Frame: Baseline to Week 156
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Number analyzed (Participants) | 201 | 213
Units on a scale | 4.1 (12.06) | 1.8 (11.79)

ADVERSE EVENTS:
Arm/Group | Carbidopa/Levodopa/Entacapone | Carbidopa/Levodopa
Serious Adverse Events (participants affected / at risk) | 91/373 | 84/371
Other Adverse Events (participants affected / at risk) | 310/373 | 291/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carbidopa/Levodopa/Entacapone (N=373) | Carbidopa/Levodopa (N=371)
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 5
Angina unstable (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac flutter (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 5 | 0
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Chalazion (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Orthostatic intolerance (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Accident at work (Injury, poisoning and procedural complications) | 1 | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Drug administration error (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 2
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0
Weight decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bursa calcification (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 5
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cartilage neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dystonia (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 2
Parkinson's disease (Nervous system disorders) | 2 | 1
Parkinsonism (Nervous system disorders) | 2 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0
Spinal claudication (Nervous system disorders) | 1 | 0
Stupor (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2
Sudden onset of sleep (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Hypersexuality (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 2
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 | 1
Stress (Psychiatric disorders) | 1 | 0
Urinary fistula (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carbidopa/Levodopa/Entacapone (N=373) | Carbidopa/Levodopa (N=371)
Constipation (Gastrointestinal disorders) | 50 | 44
Diarrhoea (Gastrointestinal disorders) | 65 | 28
Dry mouth (Gastrointestinal disorders) | 19 | 13
Dyspepsia (Gastrointestinal disorders) | 14 | 20
Nausea (Gastrointestinal disorders) | 114 | 70
Vomiting (Gastrointestinal disorders) | 22 | 9
Fatigue (General disorders) | 40 | 42
Oedema peripheral (General disorders) | 27 | 34
Bronchitis (Infections and infestations) | 20 | 20
Nasopharyngitis (Infections and infestations) | 34 | 43
Upper respiratory tract infection (Infections and infestations) | 19 | 17
Urinary tract infection (Infections and infestations) | 20 | 24
Fall (Injury, poisoning and procedural complications) | 28 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 43
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 53
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 32
Dizziness (Nervous system disorders) | 59 | 46
Dyskinesia (Nervous system disorders) | 21 | 10
Headache (Nervous system disorders) | 37 | 26
Somnolence (Nervous system disorders) | 37 | 28
Tremor (Nervous system disorders) | 11 | 26
Abnormal dreams (Psychiatric disorders) | 25 | 17
Anxiety (Psychiatric disorders) | 37 | 27
Depression (Psychiatric disorders) | 57 | 51
Insomnia (Psychiatric disorders) | 47 | 53
Rash (Skin and subcutaneous tissue disorders) | 13 | 19
Hypertension (Vascular disorders) | 19 | 27
Orthostatic hypotension (Vascular disorders) | 19 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.